CLINICAL TRIAL: NCT00593476
Title: A Pilot Study to Assess the Effects of a Pre-packaged, Portion Controlled Meal Plan on Type 2 Diabetes and Glycemic Control
Brief Title: Pilot Study to Assess Pre-packaged, Portion-controlled Meal Plan on Weight Loss
Acronym: NS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Nutrisystem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Temple U - 10854; 10854 - IRB #
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2008-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Glycemic Control; Diabetes Support and Education; Portion Control; Prepackaged meals
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCD (Active Comparator): pre-packaged, portion-controlled (PCD) meal plan for 24 weeks
  Interventions: Other: PCD
- DSE (Active Comparator): 12 weeks of diabetes support and education (DSE) (weeks 0-12) and then crosses over to 12 weeks of PCD from weeks 13-24
  Interventions: Other: DSE

INTERVENTIONS:
Other: PCD — pre-packaged, portion-controlled (PCD) meal plan for 24 weeks
  Arms: PCD
Other: DSE — 12 weeks of diabetes support and education (DSE) (weeks 0-12) and then crosses over to 12 weeks of PCD from weeks 13-24
  Arms: DSE

SUMMARY:
The purpose of this trial is to study the safety and efficacy of a pre-packaged, portion controlled meal plan on weight loss and glycemic control in overweight and obese patients with type 2 diabetes.

Aim 1 - Effects on Weight Assess the effects of a pre-packaged, portion controlled meal plan on weight loss in overweight and obese patients with type 2 diabetes.

The researchers hypothesize that the pre-packaged, portion controlled diet (PCD) will produce a greater weight loss than a diabetes support and education (DSE) program at 12 weeks. The study will be powered to detect between group differences of 3% of body weight. Secondarily, the researchers will assess whether there are any differences in weight during the secondary phase from weeks 13-24 when both groups will consume a PCD diet.

Aim 2 - Effects on Glycemic Control

Assess the effects of a pre-packaged, portion controlled meal plan on glycemic control in overweight and obese patients with type 2 diabetes.

The researchers hypothesize that the PCD will show greater improvement in HbA1c levels than a DSE group at 12 weeks. The study will be powered to detect between group differences of .5% in HbA1c. Secondarily, improvements and differences in HbA1c from weeks 13-24 when both groups are consuming a PCD will be assessed.

DETAILED DESCRIPTION:
General Design

Randomized, non-blinded, controlled clinical trial using a parallel and cross-over design of either the treatment group which receives a pre-packaged, portion-controlled (PCD) meal plan for 24 weeks (weeks 0-24) or to the control group which receives 12 weeks of diabetes support and education (DSE) (weeks 0-12) and then crosses over to 12 weeks of PCD from weeks 13-24.

Study Population

Up to 120 volunteers with type 2 diabetes who are 21-75 years of age and overweight or obese (body mass index ≥ 25 and ≤ 50 kg/m2) with a fasting HbA1c level of 6.0 or greater.

Inclusion Criteria:

Participants must meet all of the following criteria

1. Type 2 diabetic men and non-pregnant or non-lactating women between the ages of 21 to 75
2. BMI ≥ 25 and ≤ 50
3. Subjects must be willing to comply with all study-related procedures
4. Participant with screening HbA1C ≥ 6.0

Exclusion Criteria:

If participants meet one of the following criteria they will be excluded

1. Use of insulin or other pharmaceutical agent for diabetic control other than thiazolidinedione (TZD), Sulfonylurea's, or Metformin or a combination of medications.
2. BMI ≤ 24.9 or ≥ 50.1
3. Participation in another formal weight loss program within last 6 months
4. Participation in Diabetes Support and Education Program or other formal diabetes education program within last 6 months
5. Uncontrolled hypertension (systolic blood pressure > 180 or diastolic blood pressure > 100 mmHg). Participants on medication treating hypertension for at least three months are allowable.
6. Known atherosclerotic cardiovascular disease
7. History of congestive heart failure
8. History of a non-skin malignancy within the previous 5 years
9. Any major active rheumatologic, pulmonary, hepatic, renal, dermatologic disease or inflammatory condition

   Detailed Disease and Lab Value Exclusions:

   Active rheumatologic, dermatologic disease, or autoimmune/inflammatory condition will be defined as any patient who currently, or has a past medical history of chronic (> 2 weeks) immune modulating/suppressing medications.

   Active pulmonary disease will be defined as any patient who has a history of, or currently requires, daily oral corticosteroids, leukotriene inhibitors, an oxygen requirement, or ventilation support for chronic disease management.

   Active hepatic disease: defined as any patient who currently, or has a history of requiring immune modulating/suppressing medications, ammonia lowering medications, or hepatic disease related diet modifications.

   Active renal disease: defined as any patient who currently, or has a history requiring potassium phosphate lowering medications, protein restriction diet, or hemo/peritoneal dialysis.

   Lab value exclusions are limited to all routine electrolyte values outside the normal range, except glucose. (Sodium, potassium, chloride, bicarbonate, BUN, creatinine.)
10. History of testing HIV positive
11. History of alcohol or drug abuse
12. Weight-loss inducing medications or dietary supplements within 3 months prior to enrollment.
13. Weight loss > 5 kg during the last 6 months
14. Participation in any weight loss study or investigational drug study within 6 weeks prior to the screening
15. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
16. Participants with screening triglycerides above 500 mg
17. Anyone that is physically active for ≥ 30 minutes per day as assessed in clinical interview at the screening visit
18. Uncontrolled Dyslipidemia. Participants stable on medication treating dyslipidemia for at least 3 months or more is allowable.

Physical Measures

Diabetes control: Measures of HbA1c and fasting glucose will be takes at visits 1-4 to assess diabetes and glycemic control. In addition, we will track use of medications used to control diabetes.

Dyslipidemia: Lipid/lipoprotein concentrations (total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides) will be measured at visits 1-4. Current medication use will be collected at each clinic visit. We will use these data to track the incidence and prevalence of dyslipidemia.

Inflammatory Markers: Inflammation will be measured using high sensitivity C reactive protein (hs- CRP) at visits 2-4.

Electrocardiograms: Electrocardiograms will be obtained at visit 1 according to a standard protocol.

Hypertension and blood pressure measures: Through blood pressure measurements at visits 1-4, and self-reported current medication use, we will track the incidence and prevalence of hypertension as a measure of periphery artery disease.

Weight, height, and waist circumference: Body weight will be measured at each PCD visit, using calibrated scales. Participants will be weighed in light indoor clothing. Waist circumference will be measured at visits 1-4. Height will be measured at visit 1.

Serum and DNA samples: Samples of serum will be frozen and stored for future testing of new and emerging cardiovascular risk factors. DNA samples will be frozen and stored to identify genetic markers of diet response. We will use these samples to determine the possibility that the common genetic variant ENPP1 K121Q could predispose diabetic and metabolic syndrome subjects to respond better to weight loss intervention than those who have the common variant K121K. Similarly, other genetic variants that associate with obesity and insulin resistance may change susceptibility to weight loss in different directions. If at any time during the study a participant decides they do not want their serum samples to be stored they may have them destroyed

Self-Reported Measures

Psychosocial measures: A battery of psychosocial measures will be assessed including standardized assessments such as the Beck Depression Inventory8 and an eating disorders questionnaire.9 These surveys will be measured will be assessed at visits 1-4.

Quality of life: The Short Form 36 (SF-36) version will be used to measure general health related quality of life at visits 1-4.10 It can be used to calculate domain scores plus two summary scores: physical summary (four domains, 21 items), and mental health summary (four domains, 14 items).

7-day Food Records: A 7 day food record will be recorded at visits 2-4 to assess compliance with the PCD in phases 1 and 2.

Acceptability: Acceptability of each program (PCD and DSE) will be measured at visits 2-4 to determine tolerability and ease of each program.

Socio-demographics: Information on employment, household composition, and education is collected at visit 1.

Weight history, personal medical history, family medical history: At visit one only. Participants report their weights at various ages, history of weight cycling, and family and personal history of disease. Participants will be referred to appropriate treatment for any eating disorders, depression or other complications discovered as a result of the standard of care weight and lifestyle inventory and beck depression inventory administered at the screening visit. This treatment will be offered at CORE, or if participants prefer, with a provider at another location relevant to their complication.

Concomitant medications and adverse events: At visits 1-4 concomitant medications and adverse events will be recorded. Additional changes to these will be assessed as needed throughout the study.

TREATMENT

Eligible volunteers are randomly assigned to a treatment group consisting of a pre-packaged, portion controlled meal plan (PCD) or to a control group that consists of a combination diabetes support and education (DSE) program/pre-packaged, portion controlled meal plan (PCD) cross-over group. Treatment assignments are unmasked. At the end of 24 weeks the treatment group will have completed 18 group sessions and the control group will have completed 15 group sessions. The PCD program is aimed at achieving and maintaining a decrease in weight from 1-24 weeks. Combination DSE/PCD program is aimed at achieving and maintaining a decrease in weight from weeks 13-24. A Certified Diabetes Educator will review the effects of diet and weight loss, exercise, and medications on blood glucose levels among all participants at the first group meeting before any changes in dietary intake or exercise are prescribed. Participants will be counseled on strategies to prevent hypoglycemia. In addition the causes, symptoms and treatment of hypoglycemia will be reviewed including when to contact their health care provider.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria.

1. Type 2 diabetic men and non-pregnant or non-lactating women between the ages of 21 to 75
2. BMI ≥ 25 and ≤ 50
3. Subjects must be willing to comply with all study-related procedures
4. Participant with screening HbA1C ≥ 6.0

Exclusion Criteria:

If participants meet one of the following criteria they will be excluded.

1. Use of insulin or other pharmaceutical agent for diabetic control other than thiazolidinedione (TZD), Sulfonylurea's, or Metformin or a combination of medications.
2. BMI ≤ 24.9 or ≥ 50.1
3. Participation in another formal weight loss program within last 6 months
4. Participation in Diabetes Support and Education Program or other formal diabetes education program within last 6 months
5. Uncontrolled hypertension (systolic blood pressure > 180 or diastolic blood pressure > 100 mmHg). Participants on medication treating hypertension for at least three months are allowable.
6. Known atherosclerotic cardiovascular disease
7. History of congestive heart failure
8. History of a non-skin malignancy within the previous 5 years
9. Any major active rheumatologic, pulmonary, hepatic, renal, dermatologic disease or inflammatory condition

   Detailed Disease and Lab Value Exclusions:
   * Active rheumatologic, dermatologic disease, or autoimmune/inflammatory condition will be defined as any patient who currently, or has a past medical history of chronic (> 2 weeks) immune modulating/suppressing medications.
   * Active pulmonary disease will be defined as any patient who has a history of, or currently requires, daily oral corticosteroids, leukotriene inhibitors, an oxygen requirement, or ventilation support for chronic disease management.
   * Active hepatic disease: defined as any patient who currently, or has a history of requiring immune modulating/suppressing medications, ammonia lowering medications, or hepatic disease related diet modifications.
   * Active renal disease: defined as any patient who currently, or has a history requiring potassium phosphate lowering medications, protein restriction diet, or hemo/peritoneal dialysis.

   Lab value exclusions are limited to all routine electrolyte values outside the normal range, except glucose. (Sodium, potassium, chloride, bicarbonate, BUN, creatinine.)
10. History of testing HIV positive
11. History of alcohol or drug abuse
12. Weight-loss inducing medications or dietary supplements within 3 months prior to enrollment.
13. Weight loss > 5 kg during the last 6 months
14. Participation in any weight loss study or investigational drug study within 6 weeks prior to the screening
15. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
16. Participants with screening triglycerides above 500 mg
17. Anyone that is physically active for ≥ 30 minutes per day as assessed in clinical interview at the screening visit
18. Uncontrolled Dyslipidemia. Participants stable on medication treating dyslipidemia for at least 3 months or more is allowable.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Changes in weight at 12 weeks. | 12 weeks

SECONDARY OUTCOMES:
Changes in HbA1c, lipids, inflammatory markers (hs-CRP), fasting glucose, blood pressure, waist circumference and survey measures at 12 weeks. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University - Center for Obesity Research and Education
Locations (2):
- United States (2):
  - Jeanes Hospital Medical Office Building, Philadelphia, Pennsylvania
  - Center for Obesity Research and Education, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] McAndrew LM, Napolitano MA, Pogach LM, Quigley KS, Shantz KL, Vander Veur SS, Foster GD. The impact of self-monitoring of blood glucose on a behavioral weight loss intervention for patients with type 2 diabetes. Diabetes Educ. 2013 May-Jun;39(3):397-405. doi: 10.1177/0145721712449434. Epub 2012 Jun 26. PMID 22735195
- [Derived] Foster GD, Borradaile KE, Vander Veur SS, Leh Shantz K, Dilks RJ, Goldbacher EM, Oliver TL, Lagrotte CA, Homko C, Satz W. The effects of a commercially available weight loss program among obese patients with type 2 diabetes: a randomized study. Postgrad Med. 2009 Sep;121(5):113-8. doi: 10.3810/pgm.2009.09.2046. PMID 19820280